CLINICAL TRIAL: NCT01760564
Title: Application of Miglustat in Patients With Niemann-Pick Type C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200802043M
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-11

CONDITIONS: Niemann-Pick Disease Type C
Keywords: Niemann-Pick disease type C; miglustat
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miglustat (Experimental): miglustat 200mg tid
  Interventions: Drug: Miglustat

INTERVENTIONS:
Drug: Miglustat — miglustat 200mg tid for adult. For children surface area correction will be made. A lower dose may be used initially to decrease side effect.
  Other Names: Zavesca

SUMMARY:
To evaluate the changes in cognitive function after miglustat treatment in Niemann-Pick type C patients.

DETAILED DESCRIPTION:
Patients with Niemann-Pick C disease will be treated with Miglutat 200mg tid. Neurologic evaluation and safety will be monitored periodically.

ELIGIBILITY:
Inclusion Criteria:

* Confirm diagnosis of Niemann-Pick C disease
* Symptomatic including motor or mental symptoms

Exclusion Criteria:

* Unknown severe diarrhea for more than 7 day
* Allergy to miglustat

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Swallowing | 12th month
  videofluoroscopic swallowing study (VFSS), or NP-C functional disability rating scale if VFSS can not be performed due to safety issue

SECONDARY OUTCOMES:
Mental | 12th month
  IQ test or Mini-Mental Status Examination if a full IQ test can not be performed

CONTACTS AND LOCATIONS:
Overall Officials: Whu-Liang Hwu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Chien YH, Peng SF, Yang CC, Lee NC, Tsai LK, Huang AC, Su SC, Tseng CC, Hwu WL. Long-term efficacy of miglustat in paediatric patients with Niemann-Pick disease type C. J Inherit Metab Dis. 2013 Jan;36(1):129-37. doi: 10.1007/s10545-012-9479-9. Epub 2012 Apr 5. PMID 22476655